CLINICAL TRIAL: NCT05493566
Title: A Biomarker Study of Low-Dose IL-2 Plus Pembrolizumab in Patients With Stage IV Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Low-Dose Interleukin-2 and Pembrolizumab for the Treatment of Stage IV Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jennifer Carlisle, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003612; NCI-2022-00931 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00003612 (Other: Emory University Hospital/Winship Cancer Institute); WINSHIP5477-21 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2022-08-02; First posted 2022-08-09 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Lung Non-Small Cell Carcinoma; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — aldesleukin; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (pembrolizumab, aldesleukin) (Experimental): Patients will be treated with pembrolizumab 200 mg IV once every 3 weeks in combination with IL-2 given at 5 million IU subcutaneously twice daily for 3 weeks (5 days on, 2 days off each week, first dose in clinic and subsequent doses at home). IL-2 will be given only for the three weeks, after which pembrolizumab will be continued as monotherapy at either 200 mg every 3 weeks or 400 mg every 6 weeks.
  Interventions: Biological: Aldesleukin; Biological: Pembrolizumab

INTERVENTIONS:
Biological: Aldesleukin — Given SC
  Other Names: 125-L-Serine-2-133-interleukin 2; Proleukin; r-serHuIL-2; Recombinant Human IL-2; Recombinant Human Interleukin-2
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This early phase 1 trial will investigate the combination of low-dose interleukin-2 (IL-2) and pembrolizumab in patients with previously untreated stage IV non-small cell lung cancer (NSCLC). Preclinical data demonstrate reinvigoration of exhausted T cells into an effector-like phenotype with improved anti-tumor activity in response to this combination. This study will evaluate T cell function as well as clinical outcomes associated with this combination therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess phenotypic, transcriptional, and epigenetic profiles of PD-1+ CD8 T cells response in patients with stage IV non-small cell lung cancer (NSCLC) treated with the combination of IL-2 and pembrolizumab.

SECONDARY OBJECTIVE:

I. To evaluate anti-tumor activity of the combination of IL-2 and pembrolizumab by assessing the objective response rate (ORR) by Response Evaluation Criteria in Solid Tumors (RECIST 1.1).

II. To evaluate the safety of the combination of IL-2 and pembrolizumab.

OUTLINE:

Patients will be treated with pembrolizumab 200 mg IV once every 3 weeks in combination with IL-2 given at 5 million IU subcutaneously twice daily for 3 weeks (5 days on, 2 days off each week, first dose in clinic and subsequent doses at home). IL-2 will be given only for the three weeks, after which pembrolizumab will be continued as monotherapy at either 200 mg every 3 weeks or 400 mg every 6 weeks.

After completion of the study treatment, patients are followed for up for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have Stage IV non-small cell lung cancer (NSCLC), based on the 8th edition of the American Joint Committee on Cancer (AJCC) NSCLC Staging System. This includes adenocarcinoma and squamous cell carcinoma.
2. Patients must have measurable disease, as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria.
3. No prior therapy for advanced NSCLC.
4. Patients with brain metastasis are eligible if they are asymptomatic or treated and stable.
5. Age greater than or equal to 18 years.
6. Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
7. Life expectancy of greater than 12 weeks.
8. Patients must have adequate organ and marrow function, including:

   1. Absolute neutrophil count (ANC) ≥ 1,500/mcL
   2. Platelet count ≥ 100,000/mcL
   3. Hemoglobin ≥ 9.0 g/dL (patients may be transfused to meet this)
   4. Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) ≤ 2.5 x institutional upper limit of normal (ULN)
   5. Serum bilirubin l≤ 1.5 x ULN
   6. Creatinine Clearance > 60 mL/min
9. Patients must have tumor PD-L1 expression of ≥1% (by 22c3 PD-L1 companion testing); patients whose PD-L1 status could not be determined are also eligible. Patients with known PD-L1 of 0% will be excluded.
10. For women of childbearing potential or men with sexual partners of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use a contraceptive method with a failure rate of < 1% per year during the treatment period and for at least 5 months after the last dose of study treatment.

    1. A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (≥12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus).
    2. Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
11. Ability to understand and the willingness to sign a written informed consent document.

    Exclusion Criteria:

    An individual who meets any of the following criteria will be excluded from participation in this study:
12. Any prior chemotherapy or immunotherapy for advanced lung cancer.
13. Prior treatment with anti-PD-1 or anti-PD-L1 therapies or pathway-targeting agents.
14. Any targetable driver mutation (e.g. ALK, EGFR exon 19 del, etc).
15. Patients with prior allogeneic bone marrow transplantation or prior solid organ transplantation.
16. Major surgical procedure within 28 days prior to cycle 1, day 1.
17. Evidence of visceral crisis (severe organ dysfunction as assessed by signs, symptoms, and laboratory values, resulting from rapid progression of neoplastic disease).
18. Active concomitant malignancy that requires therapy.
19. Treatment with systemic immunosuppressive medications (e.g., prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 2 weeks prior to Cycle 1, Day 1.

    1. Patients who have received acute, low-dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea or premedication for contrast dye allergy) are eligible.
    2. The use of inhaled corticosteroids for chronic obstructive pulmonary disease (COPD) and mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed.
20. History or risk of autoimmune disease, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Bell's palsy, Guillain-Barré syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, or glomerulonephritis

    1. Patients with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone are eligible.
    2. Patients with controlled type 1 diabetes mellitus on a stable insulin regimen are eligible.
    3. Patients with eczema, psoriasis, or lichen simplex chronicus of vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible provided they meet the following conditions:

       * Rash must cover < 10% of body surface area (BSA)
       * Disease is well controlled at baseline and only requiring low potency topical steroids (e.g., hydrocortisone 2.5%, hydrocortisone butyrate 0.1%, fluocinolone 0.01%, desonide 0.05%, alclometasone dipropionate 0.05%)
       * No acute exacerbations of underlying condition within the last 12 months (requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, high potency or oral steroids)
21. History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest CT scan.
22. QTc of >470 msec by EKG.
23. Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis, cirrhosis, fatty liver, and inherited liver disease.
24. Known HIV infection.
25. Active tuberculosis.
26. Administration of a live, attenuated influenza vaccine (e.g., FluMist) within 4 weeks before Cycle 1, Day 1 or at any time during the study.
27. Severe infections within 4 weeks prior to Cycle 1, Day 1, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia.
28. Treatment with an investigational agent for any condition within 4 weeks prior to Cycle 1, Day 1 (or within five half-lives of the investigational product, whichever is longer).
29. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
30. Patients who are pregnant or lactating, or who are intending to become pregnant during the study.

    1. Women of childbearing potential must have a negative serum pregnancy test result within 14 days prior to initiation of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2027-01-07 (Estimated); Study Completion 2028-01-07 (Estimated)

PRIMARY OUTCOMES:
Immune Response To Combination IL-2 and Pembrolizumab | Change from Baseline at weeks 1, 2, 3, 6, 12, and 18
  Percentage of patients that express a greater than 1.5-fold increase in Ki-67 + PD-L1 + CD8 T cells in peripheral blood by week 3 of combination therapy. A 95% exact confidence interval will be estimated using the Clopper-Pearson method. Descriptive statistical analysis will be utilized to determine frequencies and percentages for categorical measurements.

SECONDARY OUTCOMES:
Objective Response Rate | Up 6 weeks after study completion
  Will be calculated as proportion (Yes/[Yes + No]) along with 95% confidence intervals using the Clopper-Pearson method. Chi-square test or Fisher's exact test will be used to compare the response rate between the different groups stratified by dose level or other factors, respectively. Logistics regression model will be further employed to test the adjusted effect of dosage on the response rate after adjusting for other clinical factors and demographic factors.
Progression Free Survival (PFS) | 6 months, 1 year, 3 year, and 5 years
  Will be estimated alone with 95% confidence interval (CI). Cox proportional hazards models will be further used in the multivariable analyses to assess adjusted effect of dose levels on the patients' PFS after adjusting for other factors.
Overall Survival (OS) | 6 months, 1 year, 3 year, and 5 years
  Will be estimated alone with 95% CI. Cox proportional hazards models will be further used in the multivariable analyses to assess adjusted effect of dose levels on the patients' OS after adjusting for other factors.
Dose-limiting Toxicities (DLTs) | Up 6 weeks after study completion
  Will be summarized descriptively, and percentage of DLTs will be reported. Tumor response, assessed using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria, will be summarized descriptively using frequencies and percentages. Paired assessments of mean expression will be compared using paired t-tests or Wilcoxon signed rank tests, where appropriate. Statistical significance will be assessed using the 0.05 level, and analysis will be performed using SAS 9.4.
Incidence of Adverse Events (AEs) | Up 6 weeks after study completion
  The number and percentage of subjects who experience AEs will be presented in tabular and/or graphical format and summarized descriptively, where appropriate. AEs will be presented with and without regard to causality based on the investigator's judgment. The frequency of overall toxicity, categorized by toxicity grades 1 through 5, will be described. Additional summaries will be provided for AEs that are observed with higher frequency.

CONTACTS AND LOCATIONS:
Overall Officials: Suresh S Ramalingam, MD, FACP, FASCO, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (1):
- Emory University/Winship Cancer Institute, Atlanta, Georgia, United States